CLINICAL TRIAL: NCT00002382
Title: An Open Label International Compassionate Treatment Program for the Use of Saquinavir (R0 31-8959) Either As Monotherapy or in Combination With Other Anti-Retroviral Drugs in Patients With Proven HIV Infection
Brief Title: A Study of Saquinavir Used Alone or in Combination With Other Anti-HIV Drugs in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 229L; SV14974
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-06

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Saquinavir; Patient Selection; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir

INTERVENTIONS:
Drug: Saquinavir

SUMMARY:
To offer an investigational agent (saquinavir) to people with HIV/AIDS who are in need of additional treatment options and are not eligible to enroll in ongoing clinical trials.

Patients who no longer benefit from existing antiretroviral therapy and who are not currently enrolled in ongoing saquinavir trials are eligible for this compassionate treatment program.

DETAILED DESCRIPTION:
Patients who no longer benefit from existing antiretroviral therapy and who are not currently enrolled in ongoing saquinavir trials are eligible for this compassionate treatment program.

Patients may be registered with the program through their physicians, who will be responsible for supervising the administration of treatment; following guidelines for saquinavir dose interruption, dose reduction, or discontinuation; and assessing patient progress throughout the duration of the study. Access to saquinavir will be determined by a lottery system; 60 percent of the program slots will be reserved for patients with CD4 counts of 50 or less and the remaining 40 percent of the slots will be devoted to patients with CD4 counts between 51 and 300.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Sero-positivity for HIV -1 antibody by an ELISA test, with confirmation by an alternative method.
* CD4 count <= 300 cells/mm3 (within 4 weeks prior to entry).
* Signed, informed consent from a parent or legal guardian for patients < 18 years of age.
* Failed previous therapy with or be intolerant to other registered anti-retroviral drugs.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Eligibility for any controlled clinical study of any experimental HIV therapy.
* Grade 4 hematologic and/or Grade 3 hematologic toxicity at baseline.

Patients with the following prior conditions are excluded:

Known hypersensitivity to saquinavir or other protease inhibitors. 1. Drugs, such as rifampin and rifabutin, which induce hepatic enzymes are likely to result in decreased levels of saquinavir and, therefore, should be avoided where possible.

* Concomitant therapy and treatment should be kept at a minimum.
* Current participation in any study formally excluding concomitant treatment with experimental drugs.

  1. Saquinavir can be used in combination with other registered anti-retroviral drugs such as ZDV, ddC and/or ddl. Other not yet registered anti-retroviral drugs can be used in combination with saquinavir when these drugs are widely available in the respective country or when they are allowed in combination treatment in any on-going clinical study.
* Prophylactic treatment for any opportunistic infections.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000

CONTACTS AND LOCATIONS:
Locations (1):
- Hoffmann - La Roche Inc, Nutley, New Jersey, United States